CLINICAL TRIAL: NCT00858195
Title: A Relative Bioavailability Study of 75mg Indomethacin Extended-Release Capsules Under Fasting Conditions
Brief Title: A Relative Bioavailability Study of 75mg Indomethacin Extended-Release Capsules
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Sandoz (Industry)
Responsible Party: Eric Mittleberg, Ph.D., VP Product Development, Sandoz Inc
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: R06-0547
Record Dates: First submitted 2009-03-05; First posted 2009-03-09 (Estimated); Last update posted 2017-03-29 (Actual); Status verified 2009-03

CONDITIONS: Inflammation
Keywords: Anti-inflammatory
MeSH Terms: conditions — Inflammation | interventions — Indomethacin

ARMS (2):
- 1 (Experimental): Indomethacin 75mg ER Capsules
  Interventions: Drug: Indomethacin 75mg Extended-Release Capsules, Sandoz
- 2 (Active Comparator): Indocin 75mg SR Capsules
  Interventions: Drug: Indocin 75mg SR Capsules

INTERVENTIONS:
Drug: Indomethacin 75mg Extended-Release Capsules, Sandoz
  Arms: 1
Drug: Indocin 75mg SR Capsules
  Arms: 2

SUMMARY:
The purpose of this study is to demonstrate the bioequivalence of Indomethacin ER Capsules.

ELIGIBILITY:
Inclusion Criteria:

* No clinically significant abnormal findings on physical exam, medical history or clinical laboratory results on screening

Exclusion Criteria:

* Positive test results for HIV or hepatitis B or C
* No allergies to indomethacin or related drugs

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 36 (Actual)
Dates: Start 2006-06; Primary Completion 2006-07 (Actual); Study Completion 2006-07 (Actual)

PRIMARY OUTCOMES:
Bioequivalence according to US FDA guidelines. | 8 days

CONTACTS AND LOCATIONS:
Overall Officials: Anthony R Godfrey, Pharm. D., Principal Investigator — PRACS Institute, LTD.